CLINICAL TRIAL: NCT01523301
Title: Double Blind, Placebo-controlled, Parallel, Multicenter, Randomized Interventional Phase IV Study to Evaluate the Efficacy of Rotigotine on Depressive Symptoms in Idiopathic Parkinson's Disease Patients
Brief Title: Rotigotine Versus Placebo to Evaluate the Efficacy on Depressive Symptoms in Idiopathic Parkinson's Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP1041
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro; Depressive Symptom; Idiopathic Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine, daily doses, treatment group
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo, daily doses, placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine — Transdermal Patch
  Content:
  2 mg /24 h (10 cm^2), 4 mg /24 h (20 cm^2), 6 mg /24 h (30 cm^2), 8 mg /24 h (40 cm^2)
  * For early-stage Parkinson's disease, Subjects received Rotigotine patches in escalating weekly dose (starting with daily doses 2 mg/24 h to 8 mg/24 h) for a maximum 4-week Titration Period, then 8 week Maintenance period
  * For advanced-stage Parkinson's disease, Subjects received Rotigotine patches in escalating weekly dose (starting with daily doses 4 mg/24 h to 16 mg/24 h) for a maximum 7-week Titration Period, then 8 week Maintenance period
  Arms: Rotigotine
Drug: Placebo — Transdermal Patch
  Size:
  10 cm^2, 20 cm^2, 30 cm^2, 40 cm^2
  Subjects randomized to placebo received matching placebo patches
  Arms: Placebo

SUMMARY:
The purpose of this study was to show superiority of Rotigotine over placebo on improvement of depressive symptoms in subjects with idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
The study included a maximum 2-week Screening Period, a maximum 4-week Titration Period for early-stage Parkinson's disease or maximum 7-week Titration Period for advanced-stage Parkinson's disease, 8-week Maintenance Period, a maximum 6-day De-escalation Period for early-stage Parkinson's disease or maximum 12-day De-escalation Period for advanced-stage Parkinson's disease and 30-day Safety Follow-Up Period.

The maximum study durations for an individual subject with early-stage Parkinson's disease and with advanced-stage Parkinson's disease were 19 weeks and 23 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 20 years old
* Subjects diagnosed with idiopathic Parkinson's disease (according to the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria for Parkinson's disease) at modified Hoehn and Yahr Scale stages I-III; do not have motor fluctuations, dyskinesia, and have stable motor symptom at least 4 weeks prior to the Screening Visit as judged by the local investigator
* Subject has a Beck Depression Inventory II (BDI-II) score ≥ 16 as evidenced by depression rating scale study in Parkinson's disease (Schrag A et al, 2007)
* Subject has a Mini-Mental State Examination (MMSE) score ≥ 24
* If subject is taking Levodopa (L-DOPA) and derivatives, Monoamine Oxidase (MAO) B-inhibitors, anticholinergics agents, Catechol-O-Methyl Transferase (COMT) inhibitor or N-Methyl-D-Aspartate (NMDA) antagonist, he/she must have been on stable dose for at least 28 days prior to the Screening Visit
* If subject is taking an antidepressant drug such as selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), bupropion, tricyclic antidepressants (TCAs), he/she must have been on a stable dose for at least 28 days prior to the Screening Visit and be maintained on that dose for the duration of the trial

Exclusion Criteria:

* Subject has any medical or psychiatric condition (ie, bipolar disorder, dementia, hallucinations or psychosis) that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the C-SSRS at Screening (Visit 1)
* Current psychotherapy or behavior therapy while participating in this study
* Subject has received electroconvulsive therapy within 12 weeks of the Screening Visit
* Subject who has received dopamine agonists within 28 days of the Screening Visit
* Subject who has received neuroleptics, methylphenidate, reserpine, alpha-methyldopa, metoclopramide, levosulpiride or amphetamine derivatives within 28 days of the Screening Visit

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (29):
- South Korea (29):
  - 03, Ansan
  - 19, Anyang
  - 08, Busan
  - 26, Busan
  - 04, Daegu
  - 05, Daegu
  - 16, Daejeon
  - 28, Goyang
  - 24, Gwangju
  - 29, Gwangju
  - 11, Gyeonggi-do
  - 15, Jinju
  - 23, Jungbuk
  - 01, Seoul
  - 02, Seoul
  - 06, Seoul
  - 07, Seoul
  - 09, Seoul
  - 10, Seoul
  - 12, Seoul
  - 13, Seoul
  - 14, Seoul
  - 17, Seoul
  - 18, Seoul
  - 20, Seoul
  - 21, Seoul
  - 22, Seoul
  - 27, Seoul
  - 25, Yangsan

REFERENCES:
- [Derived] Chung SJ, Asgharnejad M, Bauer L, Ramirez F, Jeon B. Evaluation of rotigotine transdermal patch for the treatment of depressive symptoms in patients with Parkinson's disease. Expert Opin Pharmacother. 2016 Aug;17(11):1453-61. doi: 10.1080/14656566.2016.1202917. Epub 2016 Jul 7. PMID 27322571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This double-blind, randomized, multicenter, placebo-controlled, in-Patient study started recruiting in April 2012.
Pre-assignment Details: Participant flow refers to the Randomized Set (RS), consisting of all randomized subjects.
Groups:
- Rotigotine: Rotigotine, daily doses, treatment Group.
  Early-stage Parkinon´s disease for 1 week: Rotigotine dose at 2 mg/24 h. Advanced-stage Parkinson´s disease for 1 week: Rotigotine dose at 4 mg/24 h.
  Afterwards the dose has been increased in the Titration Period by 2 mg/24 h each week until either the optimal or maximal dose was reached.
  All subjects remained 8-weeks in the Maintenance Period. In the De-escalation Period Subjects with early-stage Parkinson´s disease de-escalated their dose by 2 mg/24 h every other day to 2 mg/24h, and then to 0 mg after 2 days. Subjects with advanced-stage Parkinson´s disease de-escalated their dose by 2 mg/24h every other day to 4 mg/24h, and then to 0 mg after 2 days.
  A Safety Follow-Up Visit was scheduled for all subjects 30 days after their last dose administration.
- Placebo: Placebo, daily doses, placebo Group. Subjects randomized to placebo received matching placebo patches.
  Early-stage Parkinson´s disease for 1 week: Placebo patches´ dose at 2 mg/24 h. Advanced-stage Parkinson´s disease for 1 week: Placebo patches´dose at 4 mg/24 h.
  Afterwards the dose has been increased in the Titration Period by 2 mg/24 h each week until either the optimal or maximal dose was reached.
  All subjects remained 8-weeks in the Maintenance Period.
  In the De-escalation Period Subjects with early-stage Parkinson´s disease de-escalated their dose by 2 mg/24 h every other day to 2 mg/24h, and then to 0 mg after 2 days. Subjects with advanced-stage Parkinson´s disease de-escalated their dose by 2 mg/24h every other day to 4 mg/24h, and then to 0 mg after 2 days.
  A Safety Follow-Up Visit was scheduled for all subjects 30 days after their last dose administration.
Period: Overall Study
Arm/Group | Rotigotine | Placebo
Started | 184 | 196
Completed | 149 | 164
Not Completed | 35 | 32
Not completed — Adverse Event | 25 | 16
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Other Reason | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS), which consists of all randomized subjects.
Arm/Group | Rotigotine | Placebo | Total Title
Number analyzed (Participants) | 184 | 196 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.9) | 64.9 (8.2) | 65.2 (8.5)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  >18-<65 years | 76 | 88 | 164
  >=65 years | 108 | 108 | 216
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 122 | 218
  Male | 88 | 74 | 162
Weight [Mean (Standard Deviation); unit: kg] | 61.54 (9.68) | 62.24 (9.84) | 61.90 (9.76)
Height [Mean (Standard Deviation); unit: cm] | 160.04 (8.41) | 159.17 (8.14) | 159.59 (8.27)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of Maintenance Period in the Score of the Hamilton Depression Scale (HAM-D)
Description: The HAM-D consists of 17 items. Nine of the items are scored on a 5-point scale, ranging from 0 to 4. The remaining 8 items are scored on a 3-point scale, from 0 to 2. Therefore, the total score ranges between 0 to 52, with a cutoff score of 15/16 diagnosing major depressive disorder.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 15)
Population: Efficacy Evaluable Set (EES) consisted of all subjects from the Full Analysis Set (FAS) with a baseline total HAM-D score of 12 or larger.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Efficacy Evaluable Set (Rotigotine Treated Subjects): Rotigotine, daily doses, treatment Group. The Efficacy Evaluable Set (EES) consisted of all subjects who received at least one dose of study medication, had a valid Baseline and at least 1 valid post-Baseline HAM-D 17 measurement and who had a Baseline HAM-D 17 score of 12 or higher.
- Efficacy Evaluable Set (Placebo Treated Subjects): Placebo, daily doses, placebo Group. The Efficacy Evaluable Set (EES) consisted of all subjects who received at least one dose of study medication, had a valid Baseline and at least 1 valid post-Baseline HAM-D 17 measurement and who had a Baseline HAM-D 17 score of 12 or higher.
Arm/Group | Efficacy Evaluable Set (Rotigotine Treated Subjects) | Efficacy Evaluable Set (Placebo Treated Subjects)
Number analyzed (Participants) | 120 | 131
units on a scale | -4.79 [-5.87 to -3.71] | -3.68 [-4.68 to -2.67]
Statistical Analysis 1: Comparison: Efficacy Evaluable Set (Rotigotine Treated Subjects) vs Efficacy Evaluable Set (Placebo Treated Subjects); The change from Baseline to the end of the Maintenance period in the score of the HAM-D of rotigotine-treated subjects has been compared with those subjects on placebo in the EES. The null hypothesis (H0) was that there was no difference in the change of the HAM-D score between the active treatment and the placebo group. The alternative hypothesis (H1) was that there was a difference in the change of HAM-D score between the rotigotine and the placebo arm; Test type: Superiority or Other; p = 0.1286, ANCOVA — The null hypothesis was assessed with a 2-sided test and not rejected at p≤0.05; Difference in LS Mean = -1.12, 95% CI 2-sided [-2.56 to 0.33]

2. Secondary Outcome: Change From Baseline to the End of Maintenance Period in the Score of Beck Depression Inventory (BDI-II)
Description: The Beck Depression Inventory II (BDI-II) is a self-report instrument to measure Depression symptoms and severity. There are 21 items in the BDI-II. Scores of 0-13 are considered minimal depression; 14-19 indicates mild depression; 20-28 indicates moderate depression; and 29-63 indicates severe depression.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 15)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Efficacy Evaluable Set (Rotigotine Treated Subjects) | Efficacy Evaluable Set (Placebo Treated Subjects)
Number analyzed (Participants) | 120 | 131
units on a scale | -5.87 [-7.39 to -4.34] | -4.68 [-6.11 to -3.26]

3. Secondary Outcome: Change From Baseline to the End of Maintenance Period in the Score of Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living-ADL Subscale)
Description: The UPDRS Part II is a tool to measure Activities in Daily Living - it includes speech, salivation, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, turning in bed and adjusting clothes, falling (unrelated to freezing), freezing when walking, walking, tremor, and sensory complaints related to Parkinsonism. Each of the 13 questions is measured on a scale from 0 (normal) to 4 (severe). The total score of UPDRS part II ranges from 0 (normal) to 52 (severe).
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 15)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Efficacy Evaluable Set (Rotigotine Treated Subjects) | Efficacy Evaluable Set (Placebo Treated Subjects)
Number analyzed (Participants) | 120 | 131
units on a scale | -1.13 [-1.76 to -0.50] | -0.10 [-0.69 to 0.49]

4. Secondary Outcome: Change From Baseline to the End of Maintenance Period in the Score of Unified Parkinson's Disease Rating Scale (UPDRS) Part III (Motor Subscale)
Description: Improvement of motor symptoms is measured by the change from Baseline in UPDRS Part III motor score. The UPDRS Part III is an accepted and validated scale for the assessment of motor function in Parkinson's disease. Each of the elements in the UPDRS Part III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The total score of UPDRS part III ranges from 0 (normal) to 108 (severe abnormalities).
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 15)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Efficacy Evaluable Set (Rotigotine Treated Subjects) | Efficacy Evaluable Set (Placebo Treated Subjects)
Number analyzed (Participants) | 120 | 131
units on a scale | -3.07 [-4.28 to -1.86] | -1.65 [-2.78 to -0.52]

5. Secondary Outcome: Change From Baseline to the End of Maintenance Period in the Combined Score of Unified Parkinson's Disease Rating Scale (UPDRS) Part II (ADL) Plus Part III (Motor Subscale)
Description: The combined score of UPDRS part II and UPDRS part III is the sum of the individual scores and threfore ranges from 0 (normal) to 160 (severe).
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 15)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Efficacy Evaluable Set (Rotigotine Treated Subjects) | Efficacy Evaluable Set (Placebo Treated Subjects)
Number analyzed (Participants) | 120 | 131
units on a scale | -4.20 [-5.79 to -2.62] | -1.81 [-3.29 to -0.33]

6. Secondary Outcome: Change From Baseline to the End of Maintenance Period in the Score of Apathy Scale (AS)
Description: The AS is an abbreviated version of the Apathy Scale (AS). The AS consists of 14 items phrased as questions that are to be answered on a four-point Likert scale. It was developed specifically for patients with Parkinson Disease (PD). For questions 1-8, the scoring system is the following: not at all = 3 points; slightly = 2 points; some =1 point, a lot = 0 point. For questions 9-14: the scoring system is the following: not at all = 0 points; slightly = 1 point; some = 2 points; a lot = 3 points. Adding all scores provides the final score with a range from 0 to 42.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 15)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Efficacy Evaluable Set (Rotigotine Treated Subjects) | Efficacy Evaluable Set (Placebo Treated Subjects)
Number analyzed (Participants) | 120 | 131
units on a scale | -1.93 [-2.83 to -1.04] | -0.67 [-1.50 to 0.17]

7. Secondary Outcome: Change From Baseline to the End of Maintenance Period in the Score of Snaith-Hamilton Pleasure Scale (SHAPS)
Description: The SHAPS is a self-report instrument developed for the assessment of hedonic capacity. The sum of the 14 items scores ranges from 0 to 14. A higher score represents more anhedonic symptoms.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 15)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Efficacy Evaluable Set (Rotigotine Treated Subjects) | Efficacy Evaluable Set (Placebo Treated Subjects)
Number analyzed (Participants) | 120 | 131
units on a scale | -0.82 [-1.28 to -0.37] | -0.60 [-1.03 to -0.17]

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAE) were collected during the study, which began in April 2012 and concluded in October 2014.
Description: TEAEs are comprised of the Safety Population, which consists of all randomized subjects who received at least 1 dose of study medication.
Arm/Group | Rotigotine | Placebo
Serious Adverse Events (participants affected / at risk) | 6/184 | 14/196
Other Adverse Events (participants affected / at risk) | 112/184 | 91/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=184) | Placebo (N=196)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (4)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=184) | Placebo (N=196)
Nausea (Gastrointestinal disorders) | 42 (52) | 15 (16)
Vomiting (Gastrointestinal disorders) | 13 (14) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (12) | 10 (10)
Application site pruritus (General disorders) | 19 (20) | 10 (12)
Application site erythema (General disorders) | 11 (11) | 5 (6)
Asthenia (General disorders) | 5 (5) | 11 (13)
Nasopharyngitis (Infections and infestations) | 7 (8) | 13 (15)
Dizziness (Nervous system disorders) | 28 (31) | 25 (27)
Headache (Nervous system disorders) | 19 (22) | 20 (23)
Suicidal ideation (Psychiatric disorders) | 21 (25) | 22 (25)
Insomnia (Psychiatric disorders) | 13 (13) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (12) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.